CLINICAL TRIAL: NCT01392963
Title: The Treatment of Depression With Botulinum Type A Toxin (Botox): A Randomized, Double Blind, Crossover Study
Brief Title: The Treatment of Depression With Botulinum Type A Toxin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seton Healthcare Family (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-11-021
Record Dates: First submitted 2011-07-08; First posted 2011-07-13 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Depression
Keywords: botox; depression
MeSH Terms: conditions — Depression | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botox, Then Placebo (Experimental): At baseline visit (week 0) participants received an injection of clostridium botulinum toxin type A neurotoxin complex (Allergan; total injection of 29-40 U) in the glabella region according to standard protocols of cosmetic botulinum toxin applications. After a 3 month evaluation period, participants received a placebo injection (matching botulinum toxin) to glabella region at study visit 4 (week 12).
  Interventions: Drug: botulinum toxin type A neurotoxin complex; Drug: Placebo
- Placebo, Then Botox (Experimental): At baseline visit (week 0) participants received a placebo injection (matching botulinum toxin) to glabella region. After a 3 month evaluation period, participants received an injection of clostridium botulinum toxin type A neurotoxin complex (Allergan; total injection of 29-40 U) in the glabella region according to standard protocols of cosmetic botulinum toxin applications at study visit 4 (week 12).
  Interventions: Drug: botulinum toxin type A neurotoxin complex; Drug: Placebo

INTERVENTIONS:
Drug: botulinum toxin type A neurotoxin complex — 29-40 U injection
  Other Names: Botox, botulinum toxin type A (BTA)
Drug: Placebo — 29-40 U 0.9% NaCl injection
  Other Names: botulinum toxin type A neurotoxin complex matched injection

SUMMARY:
A 24-week Randomized, Double-blind study treating people who suffer from depression who also have moderate to severe frown lines in forehead region with Botox injections. Subjects participating will have their photos taken and complete a questionnaire regarding their depression. They will see a psychiatrist at every visit who will assess their depression.

DETAILED DESCRIPTION:
Participants will be assigned to receive either placebo or botulinum toxin injections in the forehead

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female between the ages of 18 and 65
2. Major Depression Disorder as defined by DSM IV criteria and diagnosed by a psychiatrist. DSM (Diagnostic and Statistical Manual) IV criteria for depression are: a depressed mood or anhedonia for at least a two week period. This mood must represent a change from the person's normal mood; social, occupational, educational or other important functioning must also be negatively impaired by the change in mood. Major depressive disorder cannot be diagnosed if a person has a history of bipolar disorder or if the depressed mood is better accounted for by substance abuse or a psychotic disorder. In addition, the patient must have 5 of the following symptoms:

   * Significant weight loss or weight gain.
   * Insomnia or hypersomnia
   * Psychomotor agitation or retardation
   * Feelings of worthlessness or excessive guilt
   * Poor Concentration
   * Fatigue or loss of energy
   * Suicidal thoughts
3. History of depression for at least 6 months
4. Initial score 14 or higher on initial Hamilton Depression rating scale.
5. Melancholic facial expressions amenable to treatment with Botox. Photos will be taken of potential participants and ranked independently by two investigators, on a scale of 1-10 based on how negative they look, 10 being the highest. Patients with an average score of 6 or above will be included in the study

Exclusion Criteria:

1. Active substance abuse
2. Bipolar Depression
3. Subjects who are pregnant, nursing or trying to become pregnant during study participation
4. Subjects who are currently on more than 3 psychiatric medications at the time of enrollment
5. Current medications used to treat depression must be stable for at least 60 days prior to enrollment
6. Previous Botox treatment
7. The Principle Investigator has determined that this study is not in the best interest of the subject and therefore the subject will not be enrolled.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Magid, MD, Principal Investigator — Seton Healthcare Family
Locations (1):
- Seton Mind Institute: Medical Park Tower, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Magid M, Reichenberg JS, Poth PE, Robertson HT, LaViolette AK, Kruger TH, Wollmer MA. Treatment of major depressive disorder using botulinum toxin A: a 24-week randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2014 Aug;75(8):837-44. doi: 10.4088/JCP.13m08845. PMID 24910934
- [Derived] Crowley JS, Silverstein ML, Reghunathan M, Gosman AA. Glabellar Botulinum Toxin Injection Improves Depression Scores: A Systematic Review and Meta-Analysis. Plast Reconstr Surg. 2022 Jul 1;150(1):211e-220e. doi: 10.1097/PRS.0000000000009240. Epub 2022 May 20. PMID 35588104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from local outpatient psychiatry and primary care practices, and through internet advertisements and media appearances.
Pre-assignment Details: A total of 101 were screened via telephone, 39 received a face-to-face screening interview, and 30 were enrolled in the study.
Period: Week 0 (First Intervention)
Arm/Group | Botox, Then Placebo | Placebo, Then Botox
Started | 11 | 19
Completed | 11 | 17
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Week 12 (Second Intervention)
Arm/Group | Botox, Then Placebo | Placebo, Then Botox
Started | 11 | 17
Completed | 11 | 17
Not Completed | 0 | 0
Period: Week 24 Follow-up
Arm/Group | Botox, Then Placebo | Placebo, Then Botox
Started | 11 | 17
Completed | 9 | 17
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botox, Then Placebo | Placebo, Then Botox | Total
Number analyzed (Participants) | 11 | 19 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 19 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 28
  Male | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Depression Symptoms on the Hamilton Depression Rating Scale 21 (HDRS-21) AT WEEK 6
Description: HDRS-21 is a validated, clinician-administered depression assessment scale. Possible scores range from 0 - 7 (within normal range or remission) 8-16 (mild depression) 17-23 (moderate depression) 24-52 (severe depression). Change = (Week 6 post injection score - baseline week 0 score).
  PRIMARY OUTCOME MEASURE IS THE CHANGE IN HDRS-21 SCORE AFTER WEEK 6
Time Frame: baseline and week 6
Population: Participants that completed all study visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Botox, Then Placebo: At baseline visit (week 0) participants received an injection of clostridium botulinum toxin type A neurotoxin complex (Allergan; total injection of 29-40 U) in the glabella region according to standard protocols of cosmetic botulinum toxin. After a 3 month evaluation period, participants received a placebo injection (matching botulinum toxin) to glabella region at study visit 4 (week 12).
Arm/Group | Placebo, Then Botox | Botox, Then Placebo
Number analyzed (Participants) | 19 | 11
units on a scale | -0.4 (4) | -12.7 (4)
Statistical Analysis 1: Comparison: Placebo, Then Botox vs Botox, Then Placebo; Test type: Other; p = 0.001, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline (Week 0) in Depression Symptoms on the Hamilton Depression Rating Scale 21 (HDRS-21) at Week 6 (Six Weeks Post Placebo Injection at Week 0) and Week 18 (Six Weeks Post Botox Injection at Week 12)
Description: HDRS-21 is a validated, clinician-administered depression assessment scale. Possible scores range from 0 - 7 (within normal range or remission) 8-16 (mild depression) 17-23 (moderate depression) 24-52 (severe depression). Change = (Week 6/18 score - baseline week 0 score)
  Outcome measure is the change in HDRS-21 score 6 weeks after injection with placebo (week 0) and Botox (week 12) - HDRS-21 done at week 6 and week 18.
Time Frame: Baseline (Week 0), Week 6, and Week 18
Population: 2 patients in the placebo first group dropped out at crossover and were not included in the 18 week assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo, Then Botox (Week 6); Placebo, Then Botox (Week 18): Group received placebo injection at week 0 of study followed by a Botox injection at week 12. HDRS-21 scores were done six weeks after each injection (week 6 and week 18).
Arm/Group | Placebo, Then Botox (Week 6) | Placebo, Then Botox (Week 18)
Number analyzed (Participants) | 19 | 17
units on a scale | -0.4 (3) | -8.4 (3)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Botox, Then Placebo | Placebo, Then Botox
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/19
Other Adverse Events (participants affected / at risk) | 0/11 | 0/19

LIMITATIONS AND CAVEATS:
93% of participants were female. This did not allow for statistical analysis based on gender. Although statistically significant, the sample size of this study was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes